CLINICAL TRIAL: NCT00825032
Title: Effects of Unsupported Upper Extremity Exercise Training in Patients With Chronic Obstructive Pulmonary Disease: a Randomized Clinical Trial
Brief Title: Efficacy of Arm Training in COPD Patients
Acronym: UEET-COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Villa Pineta Hospital (Other)
Collaborators: University of Modena and Reggio Emilia (Other)
Responsible Party: Prof. Enrico M. Clini, Villa Pineta Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEET0307
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2009-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary disease, chronic obstructive; Upper extremity; Exercise therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: comprehensive PR (Active Comparator): Inpatient comprehensive PR program that lasted lasted 3 weeks and included a minimum of 15 daily sessions of specific training for lower extremities, education, nutritional intervention, psychosocial intervention. It complied with the recommendation of the ATS/ERS.
  Interventions: Procedure: comprehensive PR
- 2: UEET + PR (Experimental): Experimental program consisting in additional 15 daily sessions of unsupported UEET over and above the same PR program used for control patients.
  Interventions: Procedure: UEET

INTERVENTIONS:
Procedure: comprehensive PR — Inpatient comprehensive PR program that lasted lasted 3 weeks and included a minimum of 15 daily sessions of specific training for lower extremities, education, nutritional intervention, psychosocial intervention. It complied with the recommendation of the ATS/ERS.
  Other Names: Pulmonary Rehabilitation
  Arms: 1: comprehensive PR
Procedure: UEET — Experimental program consisting of 15 additional daily sessions of unsupported UEET.
  Other Names: Upper extremity exercise training
  Arms: 2: UEET + PR

SUMMARY:
Recent guidelines on pulmonary rehabilitation (PR) recommend upper extremity exercise training (UEET) in patients with chronic obstructive pulmonary disease (COPD).

The theory supporting the inclusion of upper extremity exercise training in the pulmonary rehabilitation for these patients, is based on the profound understanding of the activity of the accessory respiratory muscles, which are competitively involved in both the support of the upper extremities during activities and the ventilation. However, a systematic review of the literature carried out by our staff reveals that the clinical trials carried out up to now to verify the effectiveness of UEET are of poor methodological quality and the investigators cannot corroborate the recommendation recently made on the basis of the results of the investigators' review.

Therefore the investigators began this randomized, parallel groups, controlled clinical trial with the purpose of determining the short-term effect of unsupported UEET on the performance of the upper extremities and on symptoms perceived during activities by patients with COPD.

DETAILED DESCRIPTION:
We recruited inpatients with stable, moderate or severe COPD referred to the PR program at the regional centre of Villa Pineta Hospital.

Patients were randomized into two groups: control and intervention. Patients randomized to the control group undertook an inpatient comprehensive PR that complied with the recommendations made by the ATS/ERS and included a minimum of 15 daily sessions of specific training for lower extremities.

Patients randomized to the intervention group undertook an experimental program consisting of 15 additional daily sessions of unsupported UEET over and above the same PR program used for control patients.

Measurements of upper extremity performance and symptoms perceived were taken in both groups at baseline (T0) and at the completion of the interventions (Tend) by one physiotherapist unaware to the patient's group allocation. To verify if the experimental training leads to long-term results on the functional arm exercise capacity, some measurements were repeated at 6-months as the latest follow-up (T6months).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD
* a degree of COPD severity equal or above grade 2 (moderate) on the basis of the GOLD classification
* clinical stability for a minimum of 4 weeks
* degree of chronic dyspnea ≥ grade 2 on the Medical Research Council Dyspnea Scale

Exclusion Criteria:

* muscular-skeletal abnormalities limiting the shoulder girdle functionality
* cognitive impairment limiting participation
* previous inclusion in UEET programmes within the last 3 years
* malignancies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
6-min. ring test (6MRT) | T0=baseline, Tend (week three) , T6months (six months after the completion of the training)

SECONDARY OUTCOMES:
ADL field test | T0=baseline, Tend (week three)
LCADL | T0=baseline, Tend (week three) , T6months (six months after the completion of the training)
MRC | T0=baseline, Tend (week three)
6MWT | T0=baseline, Tend (week three)

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Costi, Dr, Principal Investigator — University of Modena and Reggio Emilia; Enrico M Clini, Professor, Study Chair — Villa Pineta Hospital and University of Modena and Reggio Emilia
Locations (1):
- Villa Pineta Hospital, Pavullo nel Frignano, Modena, Italy

REFERENCES:
- [Background] Costi S, Di Bari M, Pillastrini P, D'Amico R, Crisafulli E, Arletti C, Fabbri LM, Clini EM. Short-term efficacy of upper-extremity exercise training in patients with chronic airway obstruction: a systematic review. Phys Ther. 2009 May;89(5):443-55. doi: 10.2522/ptj.20070368. Epub 2009 Mar 12. PMID 19282362
- [Background] Ries AL, Bauldoff GS, Carlin BW, Casaburi R, Emery CF, Mahler DA, Make B, Rochester CL, Zuwallack R, Herrerias C. Pulmonary Rehabilitation: Joint ACCP/AACVPR Evidence-Based Clinical Practice Guidelines. Chest. 2007 May;131(5 Suppl):4S-42S. doi: 10.1378/chest.06-2418. PMID 17494825
- [Derived] Costi S, Crisafulli E, Degli Antoni F, Beneventi C, Fabbri LM, Clini EM. Effects of unsupported upper extremity exercise training in patients with COPD: a randomized clinical trial. Chest. 2009 Aug;136(2):387-395. doi: 10.1378/chest.09-0165. Epub 2009 Jun 30. PMID 19567487